CLINICAL TRIAL: NCT01143727
Title: Comparison of SANTYL vs. Hydrogel in Debridement of Inflamed Diabetic Foot Ulcers
Brief Title: Enzymatic Versus (vs) Autolytic Debridement of Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 017-101-09-025
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-04

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Collagenases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Santyl
  Interventions: Drug: Santyl
- B (Active Comparator): Tegaderm Hydrogel
  Interventions: Drug: Tegaderm Hydrogel

INTERVENTIONS:
Drug: Santyl — Apply one 24-hr period sufficient to cover the wound.
  Arms: A
Drug: Tegaderm Hydrogel — Apply once 24-hr period sufficient to cover the wound.
  Arms: B

SUMMARY:
This study compares two standard methods for cleaning the surface of wounds on the feet of patients with diabetes mellitus. The question being asked is whether inflammation of the wound affects the ability of one or both of the methods to work.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent document must be read, signed, and dated by the subject or the subject's legally authorized representative before conducting any study procedures or exams. In addition, the informed consent document must be signed and dated by the individual who consents the subject before conducting the screening visit. A photocopy of the signed informed consent document must be provided to the subject, and the original signed document placed in the subject's chart.
* Of either sex, aged 18 years or older.
* A diagnosis of Diabetes Mellitus, Type I or II, requiring medication to control blood glucose levels.
* A qualifying ulcer, defined as follows:

  * Ulcer grade 1 or 2 on the Wagner Classification Scale (refer to Section 9.4.1)
  * Infection / inflammation grade 1 or 2 for wound bed inflammation (refer to Section 9.4.2)
  * Has not been treated or has not responded to treatment during the past 30 days
  * Has an apparent area ≥ 3.0 cm²
* Requires debridement of the wound bed
* Is sufficiently moist to allow collection of wound fluid using a filter paper disc
* Adequate arterial blood flow evidenced by ankle brachial index (ABI) of ≥ 0.7 and ≤ 1.1; if the ABI is greater than 1.1, then toe pressure of >50 mmHg.
* Subject must be willing to use the Darco shoe off-loading device and insole, or a comparable device, as indicated.
* Subject able to follow instructions, particularly regarding the application of test articles and dressings at home. Able to apply the test articles, or has a caregiver available to apply the test articles according to the protocol.

Exclusion Criteria:

* Contraindications or known hypersensitivity to the test articles or their components.
* Cellulitis extending >2 cm around the target ulcer, lymphangitic streaking, spread beneath the superficial fascia, deep-tissue abscess, gangrene, or infection of muscle, tendon, joint or bone.
* Target ulcer tunneling per probing and visual assessment.
* Use of systemic antibiotics or any drug listed in Section 9.1.6 of this protocol within 10 days of SCR visit.
* Concomitant illness or condition which, in the opinion of the Principal - Investigator, places the subject at risk for this study.
* The Medical Monitor may declare any subject ineligible for a valid procedural or medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint
Locations (1):
- Richard C. Galperin, DPM, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults aged 18 years and older, with Type I or II diabetes mellitus and at least one inflamed diabetic foot ulcer
Groups:
- Collagenase Santyl Ointment: Santyl
  Santyl : Applied once every 24-hr period sufficient to cover the wound.
- Control: Tegaderm Hydrogel
  Tegaderm Hydrogel : Applied once every 24-hr period sufficient to cover the wound.
Period: Overall Study
Arm/Group | Collagenase Santyl Ointment | Control
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Collagenase Santyl Ointment | Control | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 4 | 3 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 61.4 (15.3) | 58.0 (17.8) | 59.8 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Wound Appearance
Description: Weekly wound appearance as assessed by BWAT-m scores. BWAT-m scores used to determine primary efficacy consist of 8 subscales, each grade an aspect of wound status on a 1-5 scale; 1=normal intact skin; 5=least desirable. Total score=8-40. Subscales: Edges, Undermining, Necrotic Tissue Type, Necrotic Tissue Amount, Exudate Type, Exudate Amount, Skin Color Surrounding Wound, and Granulation Tissue.
Time Frame: 28 days
Population: 12 subjects initially for this exploratory study. 17 subjects enrolled to ensure 12 evaluable. Intent-to-treat used for primary inference. Missing values imputed by method of population mean (BWAT-m) and last observation carried forward (wound area).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collagenase Santyl Ointment | Control
Number analyzed (Participants) | 9 | 8
units on a scale
  Baseline | 19 (5.4) | 19 (1.8)
  Week 4 | 16.9 (7.6) | 14.5 (5.4)

2. Secondary Outcome: Percent Change in Wound Area
Time Frame: 28 days
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: percentage change from baseline area
Arm/Group | Collagenase Santyl Ointment | Control
Number analyzed (Participants) | 9 | 8
percentage change from baseline area | -69.9 (39.0) [-100 to 23] | -41.6 (105.0) [-100 to 213]

ADVERSE EVENTS:
Arm/Group | Collagenase Santyl Ointment | Control
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/8
Other Adverse Events (participants affected / at risk) | 2/9 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collagenase Santyl Ointment (N=9) | Control (N=8)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collagenase Santyl Ointment (N=9) | Control (N=8)
Oedema Peripheral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release.